CLINICAL TRIAL: NCT05481320
Title: A Phone Intervention for Family Dementia Caregivers in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Minnesota (Other); National Geriatric Hospital (Other Government); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1937464; R01AG064688 (NIH)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-12

CONDITIONS: Dementia
Keywords: dementia; family caregiving; phone intervention; non-pharmacological intervention; dementia caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The active treatment is a REACH VN phone intervention, a culturally adapted version of REACH VA, a multicomponent dementia family caregiver support intervention that includes psychoeducation, stress reduction, problem-solving, and skill-building.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH VN Phone Intervention (Experimental): A multicomponent behavioral intervention to support family caregivers of persons with dementia. The enrollment session (session 0) will be conducted face-to-face. Thereafter, participants will receive 4-6 intervention sessions by phone with either audio or video call over the course of 1-3 months. The sessions will occur every 1-2 weeks depending on the needs and availability of family caregivers.
  Interventions: Behavioral: REACH VN Phone Intervention
- Enhanced control (Placebo Comparator): A single phone session focused on education about the nature of dementia.
  Interventions: Behavioral: Enhanced Control

INTERVENTIONS:
Behavioral: REACH VN Phone Intervention — 4-6 intervention sessions delivered via phone over the course of 1-3 months.
  Arms: REACH VN Phone Intervention
Behavioral: Enhanced Control — A single phone session providing education about dementia.
  Arms: Enhanced control

SUMMARY:
This is a cluster randomized controlled trial to examine the feasibility, acceptability, and preliminary efficacy of the phone version of REACH VN, a psychosocial culturally adapted Alzheimer's family caregiving intervention, to support family caregivers of persons living with dementia in Vietnam.

DETAILED DESCRIPTION:
The objective of this study is to conduct a cluster randomized controlled trial (RCT) to examine the feasibility, acceptability, and preliminary efficacy of the phone version of REACH VN (Resources for Enhancing Alzheimer's Caregiver Health in Vietnam), a psychosocial culturally adapted Alzheimer's family caregiving intervention that will be delivered over the phone with an enhanced control as the comparison. The pilot cluster RCT will test the hypothesis that family caregivers who receive the intervention will show lower caregiver burden (primary outcome) and lower depressive/anxiety symptoms (secondary outcome) compared with those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate, a family member will need to be the identified adult (i.e., age 18 and above) who is the primary informal (i.e., unpaid family member) caregiver (i.e., the person who provides the most time day-to-day care) to an older adult (i.e., age 60 and above) with dementia living in the community. If the primary caregiver is not available to participate, an alternate family member who provides substantial care (i.e., at least 4 h/day) to an older adult with dementia will be eligible to participate.
* In addition, caregivers will need to score ≥ 6 on the Zarit Burden Interview-4 (ZBI-4).
* All participants will be living in clusters in Thach That District, a semi-rural area in Hanoi. Clusters will have a minimum of 3 participants and a maximum of 15 participants.

Exclusion Criteria:

* Caregivers with difficulties in the consent process due to cognitive impairment or severe sensory impairment (i.e., visual, hearing)
* Caregivers don't have access to phone
* Individuals who are not yet adults (i.e., infants, children, teenagers)
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Geriatric Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: cluster
Period: Overall Study
Arm/Group | REACH VN Phone Intervention | Enhanced Control
Started | 30; 5 cluster | 30; 4 cluster
Completed | 25; 5 cluster | 27; 4 cluster
Not Completed | 5; 0 cluster | 3; 0 cluster
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Care recipent passed away | 0 | 1
Not completed — Out-of-window assessment | 0 | 1
Not completed — No longer a primary caregiver | 3 | 0
Not completed — Unable to contact | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REACH VN Phone Intervention | Enhanced Control | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.5) | 54.4 (11.3) | 55.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 27 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 25 | 27 | 52
Zarit Burden Interview-6 (ZBI-6) [Mean (Standard Deviation); unit: score on a scale] — This measures caregiver burden related to caregiving before intervention. Range is 0-24. A higher score indicates a higher burden.
  score on a scale | 10.2 (3.7) | 10.6 (5.2) | 10.4 (4.5)
Patient Health Questionnaire-4 (PHQ-4) [Mean (Standard Deviation); unit: score on a scale] — This measures caregiver psychological distress before intervenion (e.g., depressive and anxiety symptoms). Range is 0-12. A higher score indicates a great level of psychological distress.
  score on a scale | 4.3 (3.4) | 4.8 (3.9) | 4.6 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Interview-6 (ZBI-6)
Description: Change in caregiver burden related to caregiving. Range is 0-24. A higher score indicates a higher burden.
Time Frame: Baseline, 3 months
Population: The analytic sample included participants who completed 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN Phone Intervention | Enhanced Control
Number analyzed (Participants) | 25 | 27
score on a scale
  Baseline | 10.2 (3.7) | 10.6 (5.2)
  3-month | 8.2 (4.3) | 11.4 (5.5)

2. Secondary Outcome: Patient Health Questionnaire-4 (PHQ-4)
Description: Change in caregiver psychological distress (e.g., depressive and anxiety symptoms). Range is 0-12. A higher score indicates a greater level of psychological distress.
Time Frame: Baseline, 3 months
Population: The analytic sample included participants who completed 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH VN Phone Intervention | Enhanced Control
Number analyzed (Participants) | 25 | 27
score on a scale
  Baseline | 4.3 (3.4) | 4.8 (3.9)
  3-month | 2.2 (2.4) | 5.3 (3.6)

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected for the duration of participation in the study (i.e., up to 3 months)
Arm/Group | REACH VN Phone Intervention | Enhanced Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT05481320/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05481320/SAP_001.pdf
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT05481320/ICF_002.pdf